CLINICAL TRIAL: NCT06148883
Title: Comparison of Early Ambulatory Monitoring Strategy Versus Electrophysiological Study Approach in the Management of Patients With New Left Bundle Branch Block After Transcatheter Aortic Valve Implantation
Brief Title: Management of Patients With New Left Bundle Branch Block After Transcatheter Aortic Valve Implantation
Acronym: MONITORTAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A02699-34
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Left Bundle-Branch Block
MeSH Terms: conditions — Bundle-Branch Block | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: This is a randomized in 2 parallel group study
Masking Description: open labelled clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrocardiogram Ambulatory Monitoring for 1 month and immediate discharge (Active Comparator): In this group, Pacemaker implantation will be decided, after discharge, on documented Electrocardiogram abnormalities obtained from the 1 month Electrocardiogram Ambulatory Monitoring.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation
- Electrocardiogram Ambulatory Monitoring for infra-hisian conduction evaluation (Experimental): In this group, Pacemaker implantation will be decided, before discharge, in case of prolonged His-Ventricular interval ≥ 70 ms.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — Transcatheter Aortic Valve Implantation is the implantation of a biological aortic valve percutaneously

SUMMARY:
The purpose of this study is to show that Electrocardiogram Ambulatory Monitoring-guided strategy is superior to ElectroPhysiological Study on the rate of alive patients with an appropriate Pacemaker implantation/non-implantation, at 12 months after randomization, in patients with New Onset Persistent Left Bundle Branch Block after Transcatheter Aortic Valve Implantation.

DETAILED DESCRIPTION:
This is a prospective, multicentric, randomized in parallel group, controlled, open labelled clinical study.

* After Transcatheter Aortic Valve Implantation, all consecutive patients presenting with new onset Left Bundle Branch Block will undergo in-hospital telemetry. In case of persistence (at least 48 hours) of a stable (i.e., no change in the last 24 hours) Left Bundle Branch Block > 150 ms, and in the absence of high grade Aortic Valve block or persistent prolonged PR interval > 240 ms, patients will be eligible for the study
* After written consent will be obtained, included patients will be randomized into two groups according to a 1:1 ratio:

  * Electrocardiogram Ambulatory Monitoring for 1 month and immediate discharge. In this group, Pacemaker implantation will be decided, after discharge, on documented Electrocardiogram abnormalities obtained from the 1 month Electrocardiogram Ambulatory Monitoring. Any other clinically relevant therapeutic decision based on Electrocardiogram Ambulatory Monitoring will be taken or
  * ElectroPhysiological Study for infra-hisian conduction evaluation. Pacemaker implantation will be decided, before discharge, in case of prolonged His-Ventricular interval ≥ 70 ms
* Patients in both groups will be followed until the end of the first year after randomization. Follow-up visits will be scheduled in person at 1 and 12 months, and through telemedicine at 3 and 6 months. Appropriateness of Pacemaker implantation/non-implantation will be evaluated at each follow-up time
* In case of any occurrence of syncope, patients will be evaluated in person, by the principal investigator of each centre, to evaluate and manage the syncope as recommended by the European Society of Cardiology guidelines.

Patients will be followed-up according to current practice.

ELIGIBILITY:
Inclusion Criteria:

Patients who are 18 years or older and undergo Transcatheter Aortic Valve Implantation :

1. Presenting with New Onset Persistent Left Bundle Branch Block, defined as a new Left Bundle Branch Block >150 ms that persists at least two days after Transcatheter Aortic Valve Implantation and is stable
2. With an anticipated life expectancy >1 year
3. Who consent to participate to the study

Exclusion Criteria:

1. During in-hospital Electrocardiogram monitoring period, immediately after Transcatheter Aortic Valve Implantation and before inclusion:

   * Documented high grade Atrio Ventricular block (Atrio Ventricular block of a degree higher than Mobitz I)
   * Persistent PR interval prolongation > 240 ms
   * Occurrence of syncope or sudden cardiac death,
   * Identification of any indisputable criteria for Pacemaker implantation
   * Definitive Pacemaker implantation
2. Prior Pacemaker or Implantable Cardiac defibrillator
3. Indication for Cardiac Resynchronization Therapy or Implantable cardiac defibrillator
4. Pre-existing Left Bundle Branch Block or Right Bundle Branch Block
5. Pre-existing PR interval prolongation > 240 ms
6. Severe or moderate dementia, evaluated before Transcatheter Aortic Valve Implantation, defined as a Mini Mental State Examination < 15
7. Pregnancy or breastfeeding patient
8. No affiliation to a social security scheme
9. Adult under legal protection (trusteeship, guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Alive status with appropriate Pacemaker implantation/non-implantation | 12 months
  The primary endpoint of this study is the alive status with appropriate Pacemaker implantation/non-implantation, at 12 months after randomization.
  * Appropriate Pacemaker non-implantation:
    - Absence of syncope or sudden cardiac death in a non-implanted patient
  * Appropriate Pacemaker implantation:
    * Documented indisputable criteria for Pacemaker implantation
    * Absence of syncope or sudden cardiac death
    * Absence of upgrading procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Timone - APHM, Marseille, France

IPD SHARING:
Plan to Share IPD: No